CLINICAL TRIAL: NCT01108783
Title: Double-blind, Randomized, Placebo-controlled, Phase III Study Comparing the Efficacy and Safety of Bilastine 20 mg Once Daily and Desloratadine 5 mg for the Treatment of Seasonal Allergic Rhinitis
Brief Title: A Phase III Efficacy Study of the Symptomatic Treatment of Seasonal Allergic Rhinitis With Bilastine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Faes Farma, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BILA 1003/RAE
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Rhinitis; Allergic; Seasonal; Hay Fever; Pollen Allergy; Pollinosis; Rhinoconjunctivitis; Sneezing; Nasal itching; Nasal Congestion; Rhinorrhea; Ocular itching; Ocular redness; Tearing
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis; Sneezing; Nasal Obstruction; Rhinorrhea; Lacerations | interventions — bilastine; desloratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bilastine (Experimental)
  Interventions: Drug: Bilastine
- Desloratadine (Active Comparator)
  Interventions: Drug: Desloratadine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bilastine — 20 mg (encapsulated) tablets QD/14 days
  Arms: Bilastine
Drug: Desloratadine — 5 mg (encapsulated) tablets QD/14 days
  Other Names: Aerius
  Arms: Desloratadine
Drug: Placebo — (encapsulated) Tablets QD/14 days
  Arms: Placebo

SUMMARY:
The objective of the study was to determine the efficacy and tolerability of 20 mg of Bilastine, compared to Desloratadine and placebo for the treatment of Seasonal Allergic Rhinitis.

DETAILED DESCRIPTION:
Pivotal, double-blind, randomized, placebo-controlled, comparative with desloratadine, parallel group, international, multicenter study.The Primary endpoint was the Change in total reflective score on the scale of symptoms associated with seasonal allergic rhinitis indicated by patients at the baseline assessment and over the 2 weeks of the study. A total of 720 patients with seasonal allergic rhinitis were enrolled. Duration of treatment was 14 days, preceded by one week (7 days) of placebo.

ELIGIBILITY:
Inclusion Criteria:

* The study disease was diagnosed on the basis of clinical criteria: Nasal symptoms (presence of nasal blockage, sneezing, nasal itching and rhinorrhea) and non-nasal symptoms (ocular itching, lacrimation, itching of ears and/or palate and ocular redness), as well as the skin prick test performed at the time of selection or within the year prior to entering.
* Patients with history of Seasonal Allergic Rhinitis, positive skin prick test and symptoms were included if they were between 12 and 70 years old, gave their informed consent, attended the required visits scheduled and also underwent a complete medical examination..

Exclusion Criteria:

* Patients were excluded if they had a significant nasal abnormality which could interfere with the aim of the study, acute or chronic sinusitis, asthma or any condition, disease or hypersensitivity that could be harmed.
* Patients were not allowed to take forbidden medications or not comply the study requirements.
* Patients who were currently participating in or had participated in another clinical trial within the previous three months or were planning to travel outside of the study area during the course of the study were excluded.
* Pregnant or breast-feeding women were also excluded.
* Women of childbearing potential had a pregnancy test done

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2003-04; Primary Completion 2003-08 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
AUC of TSS | 14 days
  The area under curve (AUC) of the total symptom score (TSS) since basal visit to D14 visit according to the patient's assessment.

SECONDARY OUTCOMES:
Change in TSS. Reflective symptoms | 14 days
  Change in the reflective total score on symptom scale on D14 visit and day7 visit versus D0 visit (baseline) according to the patient´s assessment on the previous 12 hours.
Change in TSS. Instantaneous score | 14 days
  Change in the total score on symptom scale on D7 and D14 visits versus D0 visit (baseline) according to the patient's assessment (instantaneous score).
Change in total nasal symptom score (TNSS) | 14 days
  Change in nasal symptom score on symptom scale on D7 and D14 visits versus D0 visit (baseline) according to the patient's and investigator's assessment.
Change in total non-nasal symptom score (TNNSS) | 14 days
  Change in non-nasal symptom score on symptom scale on D7 and D14 visits versus D0 visit (baseline) according to the patient's and investigator's assessment
VAS of discomfort | 14 days
  Overall assessment of discomfort caused by allergic rhinitis using a visual analog scale (VAS) on D7 and D14 versus D0.
CGI | 14 days
  Investigator's overall clinical impression (CGI)
Allergic rhinitis (AR) quality of life (QoL) questionnaire | 14 days
  Quality of Life change versus baseline.
Onset of action | 2 days
  Symptoms assessment in the first 48 hours since the beginning of the treatment
Safety assessment | 14 days
  comparison of the adverse event profiles throughout the course of the study, ECGs and safety blood tests on D0 and D14.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kuna, Prof. Dr., Principal Investigator — Barlicki University Hospital, Medical University of Lodz (Poland)

REFERENCES:
- [Result] Bachert C, Kuna P, Sanquer F, Ivan P, Dimitrov V, Gorina MM, van de Heyning P, Loureiro A; Bilastine International Working Group. Comparison of the efficacy and safety of bilastine 20 mg vs desloratadine 5 mg in seasonal allergic rhinitis patients. Allergy. 2009 Jan;64(1):158-65. doi: 10.1111/j.1398-9995.2008.01813.x. PMID 19132976